CLINICAL TRIAL: NCT03344588
Title: The Role of Artery-Preserving Varicocelectomy in Subfertile Men With Severe Oligozoospermia; A Randomized Controlled Study
Brief Title: The Role of Artery-Preserving Varicocelectomy in Subfertile Men With Severe Oligozoospermia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Zahran, MD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: varicocelectomy
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Infertility, Male; Oligozoospermia; Varicocelectomy
MeSH Terms: conditions — Infertility, Male; Oligospermia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients accept to participate have to sign a written informed consent and will be unaware of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artery preserving varicocelectomy (Active Comparator): In all patients, sub-inguinal varicocelectomy will be carried out under spinal anesthesia, by a single surgeon (KS), using surgical microscope. A 2-3 cm pre-pubic incision will be performed. The cord will be grasped with a Babcock clamp and isolated over a vessel tape. Any external cremastric veins will be identified and ligated using vicryl 3/0. After opening the spermatic fascia, the vassal compartment including the vasal, cremasteric arteries and lymphatics will be separated from the pampiniform plexus compartment and preserved. In group A (APV), testicular arteries will be spared with aid of by intraoperative Doppler US (VTI intraoperative Doppler system 20 MHz). The arteries will be carefully dissected by a micro-dissector, separated over a vessel loupe, and then the remaining veins will be ligated using vicryl 3/0.
  Interventions: Procedure: artery preserving varicocelectomy
- artery ligation varicocelectomy (Active Comparator): In all patients, sub-inguinal varicocelectomy will be carried out under spinal anesthesia, by a single surgeon (KS), using surgical microscope. A 2-3 cm pre-pubic incision will be performed. The cord will be grasped with a Babcock clamp and isolated over a vessel tape. Any external cremastric veins will be identified and ligated using vicryl 3/0. After opening the spermatic fascia, the vassal compartment including the vasal, cremasteric arteries and lymphatics will be separated from the pampiniform plexus compartment and preserved. In group B (ALV), all vascular channels will be ligated without identifying or sparing the internal spermatic arteries
  Interventions: Procedure: artery ligation varicocelectomy

INTERVENTIONS:
Procedure: artery preserving varicocelectomy — During sub-inguinal varicocelectomy, testicular arteries will be spared with aid of by intraoperative Doppler US (VTI intraoperative Doppler system 20 MHz). The arteries will be carefully dissected by a micro-dissector, separated over a vessel loupe, and then the remaining veins will be ligated using vicryl 3/0.
  Arms: artery preserving varicocelectomy
Procedure: artery ligation varicocelectomy — During sub-inguinal varicocelectomy, all vascular channels will be ligated without identifying or sparing the internal spermatic arteries.
  Arms: artery ligation varicocelectomy

SUMMARY:
A male factor is responsible for almost half the cases of subfertility. Varicocele is a major cause of impaired spermatogenesis and potentially a correctable cause. It affects up to 40% of men with primary subfertility and 80% of men with secondary subfertility. Varicocelectomy is now accepted as a cost effective treatment in subfertile men with clinically palpable varicocele and impaired semen parameters. Recently, Varicocelectomy is reported to improve fertility potential in patients with severe oligozoospermia. In one such study, Varicocelectomy was associated with a statistically significant increase in sperm density and motility. Spontaneous pregnancy was achieved in16.7% of cases. In a recent meta-analysis, Varicocelectomy in men with severe oligozoospermia showed a strong trend toward improvement in pregnancy rate (PR) [OR= 1.69, 95% CI (0.951, 3.020), p= 0.073] and statistically significant increase in live birth rate (LBR)[OR=1.699, 95%CI (1.020, 2.831), p= 0.04].

The impact of ligation of internal spermatic artery (ISA) during Varicocelectomy is a matter of debate. Conventional view is arterial ligation can negatively affect testicular function and decrease the likelihood of post-operative paternity. Other investigators reported that ligation of ISA was not associated with significant changes in postoperative semen parameters, testicular size or PR in comparison to artery preservation. Moreover, laparoscopic artery-ligating Varicocelectomy was proved to be superior in the form of shorter operative time and lower recurrence rates with no difference in semen parameters or PR in comparison to laparoscopic artery-preservation varicocelectomy.

Also, isolation of ISA is not an easy task during subinguinal Varicocelectomy due to compression by external oblique aponeurosis and its inherent anatomical variation. In 29 % and 57% of the cases, the ISA is surrounded by the varicose vessels and adherent to the veins respectively. Thus, the ISA is liable to a substantial risk of accidental ligation during subinguinal Varicocelectomy.

Whether or not ligation of the ISA has a deleterious effect on the fertility outcomes in patients with severe oligozoospermia; this is not clear in the literature. This prospective randomized study was conducted to assess the impact of ISA ligation during subinguinal Varicocelectomy on fertility outcome in patients with severe oligozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* adult sub-fertile male
* with clinical varicocele (grade 2,3) severe oligozoospermia (<5 million/ml)

Exclusion Criteria:

* patients' age < 18 years, recurrent varicocele, sperm concentration >5 million/ml, history of previous inguinal surgery, concomitant female factor subfertility and refusal to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the study included males with primary infertility
Enrollment: 330 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
semen parameters changes, sperm density | at 6 months
  number/ml according to WHO criteria)
sperm motility | at 6 months
  percentage ( according to WHO criteria)

SECONDARY OUTCOMES:
clinical pregnancy rate | 1 year
  number of pregnancy in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No